CLINICAL TRIAL: NCT03594357
Title: The Relationship of Cognitive Functions to Physical and Personal Factors in Patients With Multiple Sclerosis
Brief Title: Cognitive Functions in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, research assistant, Gazi University
Other Study IDs: 437
Record Dates: First submitted 2018-07-09; First posted 2018-07-20 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Balance; Cognition; Functional exercise capacity; Fatigue; Sleep quality
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple sclerosis: MS patients (EDSS: 0-5,5)
- Control: Healthy individuals without chronic disease

SUMMARY:
Approximately 65% of multiple sclerosis (MS) patients appear to have problems in their cognitive function. Long-term memory is one of the most frequently affected functions in MS patients. Many factors play a role in the deterioration of cognitive functions because of many symptoms of MS.

The aim of this study is to investigate the relationship of cognitive function with physical factors such as balance, functional exercise capacity and personal factors such as fatigue level, mood, sleep quality in patients with MS.

DETAILED DESCRIPTION:
Patients with MS between 0-5,5 score according to the Extended Disability Status Scale (EDSS) and healthy individuals of similar age and sex to patients will be included in the study. The cognitive function, balance, functional exercise capacity, fatigue, mood, sleep quality will be evaluated once.

Investigators will use descriptive statistics and t-tests to compare variables between groups. Investigators will examine the correlations between variables using Pearson bivariate correlations. The significance level is set at p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* Participants who 18-65 years of age
* MS patients who are ambulatory (Expanded Disability Status Scale score ≤ 5,5 ) in a stable phase of the disease, without relapses in the last 3 month.

Exclusion Criteria:

* Participants who have orthopedic, vision, hearing, or perception problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MS patients who apply to the Neurological Rehabilitation Unit of Gazi University Faculty of Health Sciences will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
cognitive function | baseline
  The Brief Repeatable Battery of Neuropsychological Tests will be used. The Brief Repeatable Battery of Neuropsychological Tests (BRB-N) consists of the selective reminding, 10/36 spatial recall, symbol digit modalities, paced auditory serial addition (PASAT) and word list generation tests.

SECONDARY OUTCOMES:
Balance | baseline
  The posturography (Biodex Balance System-BioSwayTM) will be used to assess postural sway and sensory interaction. The participants will be asked to stand on both feet for 30 seconds under altered sensory conditions. The four conditions are as follows: 1. Eyes open-firm surface, 2. Eyes closed-firm surface; 3. Eyes open-foam surface, 4. Eyes closed-foam surface. Each test was repeated 3 times and the overall score was recorded.
Functional exercise capacity. | baseline
  The Six-Minute Walking Test (6-MWT) will be performed to determine the functional exercise capacity. The heart rate, blood pressure and fatigue severity of the participants are recorded before and after the test. The heart rate is assessed by a heart rate monitor and fatigue severity is assessed by the Modified Borg Scale. The participants are asked to walk as far as possible for 6 minutes in a 30-meter corridor. Finally, the walking distance will be recorded in meters.
Fatigue | baseline
  Fatigue impact scale will be used to assess fatigue. There are 40 items, each of which is scored 0 (no problem) to 4 (extreme problem), providing a continuous scale of 0-160. It is composed of three subscales that describe how fatigue impacts upon cognitive (10 items), physical (10 items) and psychosocial functioning (10 items). Cognitive functioning concerns concentration, memory, thinking and organization of thoughts. Physical functioning reflects motivation, effort, stamina and coordination. Psychosocial functioning describes the impact of fatigue upon isolation, emotions, workload and coping.A higher score indicates a higher fatigue impact.
Mood | baseline
  Beck's Depression Inventory will be used to assess mood. The 21-item self-administered survey is scored on a scale of 0-3 in a list of four statements arranged in increasing severity about a particular symptom of depression. The highest possible total for the whole test would be sixty-three. A higher score indicates a higher depression.
Sleep Quality | baseline
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. A total score of "5" or greater is indicative of poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rao SM, Leo GJ, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. I. Frequency, patterns, and prediction. Neurology. 1991 May;41(5):685-91. doi: 10.1212/wnl.41.5.685. PMID 2027484
- [Background] Rao SM, Grafman J, DiGuilio D, et al. Memory dysfunction in multiple sclerosis: its relation toworking memory, semantic encoding and implicit learning.Neuropsychology 1993; 7:364-374
- [Background] Amato MP, Zipoli V, Portaccio E. Multiple sclerosis-related cognitive changes: a review of cross-sectional and longitudinal studies. J Neurol Sci. 2006 Jun 15;245(1-2):41-6. doi: 10.1016/j.jns.2005.08.019. Epub 2006 Apr 27. PMID 16643953
- [Background] Lynch SG, Parmenter BA, Denney DR. The association between cognitive impairment and physical disability in multiple sclerosis. Mult Scler. 2005 Aug;11(4):469-76. doi: 10.1191/1352458505ms1182oa. PMID 16042232
- [Background] Sandroff BM, Pilutti LA, Benedict RH, Motl RW. Association between physical fitness and cognitive function in multiple sclerosis: does disability status matter? Neurorehabil Neural Repair. 2015 Mar-Apr;29(3):214-23. doi: 10.1177/1545968314541331. Epub 2014 Jul 8. PMID 25009224